CLINICAL TRIAL: NCT01306565
Title: Comparison Between Effect of High Dose and Low Dose of Atorvastatin in Reduction Level of CRP in Patients With Unstable Angina and NSTEMI (Non ST Elevation MI)
Brief Title: High Dose and Low Dose of Atorvastatin in Patients With Unstable Angina and NSTEMI (Non ST Elevation MI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hormozgan University of Medical Sciences (Other)
Responsible Party: Vahid Vahdatkhah, Hormozgan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Atorvastatin and CRP level
Record Dates: First submitted 2011-03-01; First posted 2011-03-02 (Estimated); Last update posted 2011-03-02 (Estimated); Status verified 2008-11

CONDITIONS: Cardiovascular Disease
Keywords: Unstable angina; NSTMI; Statin; Atorvastatin
MeSH Terms: conditions — Cardiovascular Diseases; Angina, Unstable | interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- High dose atorvastatin (Active Comparator): Three 80mg daily doses of atorvastatin
  Interventions: Drug: Low dose Atorvastatin
- Low dose Atorvastatin (Experimental): 80mg atorvastatin followed by two 20mg daily atorvastatin
  Interventions: Drug: High dose atorvastatin

INTERVENTIONS:
Drug: Low dose Atorvastatin — 80mg atorvastatin followed by two 20mg daily atorvastatin
  Other Names: Lipitor
  Arms: High dose atorvastatin
Drug: High dose atorvastatin — 80mg daily atorvastatin for 72 hours
  Other Names: Lipitor
  Arms: Low dose Atorvastatin

SUMMARY:
The aim of this study is to compare the effect of high dose and low dose of Atorvastatin in reduction level of C-reactive protein (CRP) in patients with unstable angina and NSTEMI (Non ST Elevation MI) attending Shahid Mohammadi hospital in Bandar Abbas.

DETAILED DESCRIPTION:
This study compare the effect of 80mg atorvastatin followed by two 20mg daily atorvastatin with three 80mg daily atorvastatin in reduction of CRP in patients with unstable angina and NSTEMI (Non ST Elevation MI) attending Shahid Mohammadi hospital in Bandar Abbas in 2009.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unstable angina with chest discomfort at rest with normal EKG or St depression (at least 0.1mv) in two consecutive leads or new and deep T inversion (at least 0.2mv)

Exclusion Criteria:

* Myocardial Infarction with ST elevation
* Diabetes Mellitus
* Previous statin use
* Current infectious disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
CRP reduction | 72 hours
  CRP reduction will be compared between two study groups

SECONDARY OUTCOMES:
Drug side effects | 72 hours
  Headache, Myopathy

CONTACTS AND LOCATIONS:
Overall Officials: Vahid Vahdatkhah, Principal Investigator — Hormozgan University of Medical Sciences
Locations (1):
- Hormozgan University of Medical Sciences, Bandar Abbas, Hormozgan, Iran